CLINICAL TRIAL: NCT04210258
Title: Open Label Multicenter Evaluator-blinded Post-market Clinical Follow-up (PMCF) Study to Confirm Performance and Safety of Etermis 3 and 4 in the Treatment of Moderate and Severe Wrinkles/Folds as Well as Facial Volume Enhancement
Brief Title: Post-Market Clinical Follow-up Performance and Safety Study of Etermis 3 and 4 in the Face
Acronym: POMET
Status: Completed | Type: Observational
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: M900991001
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Correction of Facial Wrinkles/Folds; Facial Volume Enhancement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Etermis 3 — Cross-linked hyaluronic dermal filler. Treatment and follow-up according to standard of care and instruction of use for filling facial moderate wrinkles (marionette lines) and/or to increase lip volume
Device: Etermis 4 — Cross-linked hyaluronic dermal filler. Treatment and follow-up according to standard of care and instruction of use for filling deep and severe volume loss (nasolabial folds and/or marionette lines) and/or to increase lip volume

SUMMARY:
To confirm the clinical performance of Etermis 3 and Etermis 4 based on the blinded investigator´s assessments on the respective Merz Aesthetics Scales from day 0 (D0) pre-injection to month 6/7 (depending on touch up) visit for nasolabial folds and marionette lines and from D0 pre-injection to month 3/4 (depending on touch up) visit for upper and lower lip fullness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects seeking hyaluronic acid dermal filler treatment to redefine/volumize/correct at least two of the indicated facial areas:

  * Nasolabial folds
  * Marionette lines
  * Upper and lower lip fullness

Exclusion Criteria:

* Subjects that have already been injected with non-resorbable filler, or that have recently been treated with any dermal filler in the region to be treated in the study
* Subjects with known sensitivity to hyaluronic acid-based products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy male and female subjects seeking hyaluronic acid dermal filler treatment to redefine/volumize/correct at least two of the indicated facial areas (NLFs, marionette lines, upper and lower lips)
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Responder rate for marionette lines after treatment with Etermis 3 based on the blinded Investigator's opinion on the Merz Aesthetics Scale "Marionette lines- At Rest" | Baseline to month 6-7
Responder rate for lips after treatment with Etermis 3 based on the blinded Investigator's opinion on the Merz Aesthetics Scale "Upper and lower lip fullness - At Rest" | Baseline to month 3-4
Responder rate for NLFs after treatment with Etermis 4 based on the blinded Investigator's opinion on the Merz Aesthetics Scale "Nasolabial folds- At Rest" | Baseline to month 6-7
Responder rate for marionette lines after treatment with Etermis 4 based on the blinded Investigator's opinion on the Merz Aesthetics Scale "Marionette lines- At Rest" | Baseline to month 6-7
Responder rate for lips after treatment with Etermis 4 based on the blinded Investigator's opinion on the Merz Aesthetics Scale "Upper and lower lip fullness - At Rest" | Baseline to month 3-4

SECONDARY OUTCOMES:
Change of blinded Investigator's assessment of marionette lines, per product from D0 pre-injection to M1 visit (before touch-up), to M2, to M3/M4, to M6/M7, to M9/M10, and to M12/M13 according to the Merz Aesthetics Scale "Marionette lines - At Rest | Baseline up to month 12-13
Change of blinded Investigator's assessment of lip volume, per product from D0 pre-injection to M1 visit (before touch-up), to M2, to M3/M4, to M6/M7, to M9/M10, and to M12/M13 according to Merz Aesthetics Scale "Upper and Lower lip fullness - At Rest" | Baseline up to month 12-13
Change of blinded Investigator's assessment of nasolabial folds, per product from D0 pre-injection to M1 visit (before touch-up), to M2, to M3/M4, to M6/M7, to M9/M10, and to M12/M13 according to the Merz Aesthetics Scale "Nasolabial folds - At Rest" | Baseline up to month 12-13
Subject's satisfaction on the global impression of changes scale (GICS) from D0 pre-injection photos to M1 visit pre-optional touch-ups, M2 visit if applicable, M3/M4, M6/M7 visit, M9/M10 visit and to M12/M13 visit. | Baseline up to month 12-13
Blinded Investigator's global opinion on clinical performance on the global aesthetic improvement scale (GAIS) from D0 pre-injection photos to M1 visit pre-optional touch-ups, M2 visit if applicable, M3/M4, M6/M7 visit, M9/M10 visit and to M12/M13 visit. | Baseline up to month 12-13

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (6):
- Germany (6):
  - Merz Investigational Site #0490099, Darmstadt
  - Merz Investigational Site #0490095, Hamburg
  - Merz Investigational Site #0490345, Hamburg
  - Merz Investigational Site #0490309, Kassel
  - Merz Investigational Site #0490368, München
  - Merz Investigational Site #0490362, Potsdam

IPD SHARING:
Plan to Share IPD: No